CLINICAL TRIAL: NCT03244761
Title: Physiological Effects of High-Flow Tracheal Oxygen Via An Modified Interface in Tracheostomized Patients
Brief Title: Physiological Effects of High-Flow Tracheal Oxygen Via An Modified Interface
Status: Completed | Type: Observational
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Jian-Xin Zhou, Professor, Capital Medical University
Other Study IDs: KY-2017-CC-13
Record Dates: First submitted 2017-08-07; First posted 2017-08-10 (Actual); Last update posted 2018-02-12 (Actual); Status verified 2017-08

CONDITIONS: Tracheostomy
Keywords: high flow tracheal oxygen; modified interface

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- The standard HFT: The high-flow oxygen was delivered via tracheostomy using a standard HFT.
- The modified HFT: The high-flow oxygen was delivered via tracheostomy using a modified HFT.
  Interventions: Procedure: The modified HFT

INTERVENTIONS:
Procedure: The modified HFT — The HFT was modified by increasing the expiratory resistance.
  Groups: The modified HFT

SUMMARY:
Tracheostomy is often performed in patients after or anticipated prolonged mechanical ventilation, who are usually required oxygen therapy after discontinuation of mechanical ventilation.

DETAILED DESCRIPTION:
Tracheostomy is often performed in patients after or anticipated prolonged mechanical ventilation, who are usually required oxygen therapy after discontinuation of mechanical ventilation.The high-flow tracheal (HFT) oxygen therapy in tracheostomized patients has been shown that can improve oxygenation,but can not induce positive end-expiratory pressure and elevation of end-expiratory lung volume. A modified HFT system by increasing expiratory resistance might induce PEEP and consequently elevate EELV.

ELIGIBILITY:
Inclusion Criteria:

* The tracheostomized patient requiring the convenient oxygen therapy.

Exclusion Criteria:

* Under 18 years;
* history of esophageal, gastric or lung surgery;
* The contraindication of using EIT (pacemaker, defibrillator, and implantable pumps).

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The tracheostomized patient
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2017-09-15 (Actual); Study Completion 2018-02-05 (Actual)

PRIMARY OUTCOMES:
The mean end expiratory pressure. | the last 1 minutes of steady breathing during the standard or modified HFT.
  The patients was delivering the high flow oxygen via the standard and modified HFT interface for 20 minutes.

SECONDARY OUTCOMES:
Changes in global and regional EELV | the last 1 minutes of steady breathing during the standard or modified HFT.
  The Electrical impedance tomography (EIT) was applied in monitoring the change of EELV at the bedside.

CONTACTS AND LOCATIONS:
Overall Officials: Jian-Xin Zhou, MD, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Jian-Xin Zhou, Beijing, Beijing Municipality, China